CLINICAL TRIAL: NCT05132777
Title: A Phase II, Open Label, Multi-center Study to Assess the Efficacy and Safety of JMT101 Combined With Osimertinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutations
Brief Title: Efficacy and Safety of JMT101 Combined With Osimertinib in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-CSP-003
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer; EGFR Exon20 Insertion Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JMT101 in combination with Osimertinib (Experimental)
  Interventions: Drug: JMT101; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: JMT101 — JMT101, 6 mg/kg, IV infusion once every two weeks (one treatment cycle is 4 weeks).
Drug: Osimertinib Mesylate Tablets — Osimertinib, 160 mg, Oral administration once daily (one treatment cycle is 4 weeks).

SUMMARY:
This study is a phase II, open label, multi-center study to evaluate the efficacy and safety of JMT101 combined with Osimertinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR exon 20 insertion mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Patients with non-irradiable, non-operable, histologically or cytologically confirmed Stage IIIB~IV NSCLC, harboring an EGFR exon 20 insertion mutation (including duplication mutations), who have progressed on or intolerable to prior platinum-based chemotherapy.
3. At least 1 measurable lesion according to RECIST 1.1.
4. ECOG score 0 or 1.
5. Life expectancy≥3 months.
6. Adequate organ function(tested within 7 days prior to the first dose): Absolute neutrophil count (ANC)≥1.5×10^9 /L, Platelets≥90×10^9/L, Hemoglobin≥9 g/dL or ≥5.6 mmol/L; Serum creatinine <1.5 × ULN; Total bilirubin ≤1.5×ULN (if liver metastases are present,≤3×ULN), AST and ALT≤3×ULN (if liver metastases are present,≤5×ULN)；INR or PT≤1.5×ULN, APTT≤1.5×ULN.
7. A female of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose. Any male and female patient of childbearing potential must agree to use effective contraception method throughout the trial period and for another half year after the end of the trial.
8. Fully understand and fully informed of this study; must sign and give the written Informed Consent Form (ICF).

Exclusion Criteria:

1. Previously received monoclonal antibody therapy targeting EGFR.
2. Previous chemotherapy, biotherapy, targeted therapy, immunotherapy or other anti-tumor treatment within 4 weeks prior to the first dose of the study drug, 2 weeks (or 5 half-lives whichever is longer) for using small molecule targeted drugs, 2 weeks for using radiotherapy..
3. Treated with other investigational agents within 4 weeks prior to the first dose of the study drug.
4. Experienced any major surgery (excluding puncture biopsy) or significant trauma within 4 weeks prior to the first dose.
5. Hypersensitivity or intolerance to our study drug or any excipients of the study drug.
6. Received strong or moderate inducers of CYP3A4 within 14 days prior to the first dose.
7. The adverse reactions of previous antitumor treatment have not yet recovered to Grade≤ 1 based on CTCAE 5.0 or baseline (except for the toxicity without safety risk judged by the investigator, such as alopecia).
8. Had untreated central nervous system metastasis or meningeal metastasis.
9. History of autoimmune disease, immunodeficiency, including HIV positive, or the presence of other acquired or congenital immunodeficiency, or organ transplantation.
10. Active hepatitis B, hepatitis C virus or syphilis infection.
11. History of severe cardiovascular disease.
12. Have difficulty with swallowing medications, or there is a condition seriously affecting the gastrointestinal absorption as judged by investigators.
13. Other malignant tumors diagnosed within 5 years prior to the first dose, with the exception of adequately treated skin basal cell carcinoma, skin squamous cell carcinoma, preinvasive cervical carcinoma or breast cancer that was effectively removed and not requiring or not expected to require other treatment during the study period.
14. History of interstitial lung disease, drug-induced interstitial lung disease, radioactive pneumonia requiring steroid treatment, or any evidence of clinical active interstitial lung disease.
15. History of other serious systemic diseases, in the judgment of the investigator, that make the subject unfit for the study.
16. Alcohol or drug dependence.
17. Had an unequivocal history of neurological or psychiatric disorders, including epilepsy or dementia.
18. Pregnant or lactating woman.
19. Not suitable for this study as determined by the investigator due to other reasons.
20. Patients harboring EGFR exon20 insertion mutation and also have other EGFR TKI-sensitizing EGFR mutations, such as G719X mutation in exon 18, exon 19 deletion mutation (19 del), exon 20 T790M or S768I mutation, exon 21 L858R mutation, or L861Q mutation.
21. Previously received drugs that developed for EGFR exon20 insertion mutated NSCLC ( such as TAK-788, Poziotinib, DZD9008 or JNJ-61186372); the short-term use is allowed, such as≤2 weeks. Responsive to previous EGFR-TKI treatment (including the best overall response of complete response, partial response, or stable disease last more than 6 months). Previously received PD-1 or PD-L1 monoclonal antibody therapy within 3 months prior to the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) Assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1 | From the first dose to disease progression or end of study, an average of 1 year

SECONDARY OUTCOMES:
Confirmed ORR Assessed by the Investigator per RECIST Version 1.1 | From the first dose to disease progression or end of study, an average of 1 year
Duration of Response (DoR) | From the first dose to disease progression or end of study, an average of 1 year
Disease control rate (DCR) | From the first dose to disease progression or end of study, an average of 1 year
Progression free survival (PFS) | From the first dose to disease progression or end of study, an average of 1 year
Overall survival (OS) | From the first dose to death or end of study, an average of 1.5 years
Incidence of adverse events (defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAEV5.0)) | From the enrollment until 30 days after the last dose
Immunogenicity profile of JMT101 | From the enrollment until 30 days after the last dose
  Blood samples will be collected at specified timepoints to detect the presence of anti-drug antibodies and neutralizing antibodies against JMT101
Area under the concentration curve from time 0 to the concentration at last time point (AUC0-last) of JMT101. | From the first dose to cycle 3 day 1 (each cycle is 28 days)
Maximum measured plasma concentration (Cmax) of JMT101. | From the first dose to cycle 3 day 1 (each cycle is 28 days)
Time to maximum plasma concentration (Tmax) of JMT101. | From the first dose to cycle 3 day 1 (each cycle is 28 days)
Half-life (T1/2) of JMT101. | From the first dose to cycle 3 day 1 (each cycle is 28 days)
Cl/F of JMT101. | From the first dose to cycle 3 day 1 (each cycle is 28 days)
Detection of cancer-related biomarkers in circulating tumor DNA from plasma to analyse the corcorrelation with clinical efficacy and drug resistance. | From the enrollment to disease progression, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No